CLINICAL TRIAL: NCT02740088
Title: Clinical Value of 18F-sodium Fluoride Uptake at the Aortic Valve for Prediction of the Progression in Patients With Moderate Aortic Stenosis: a Prospective Study
Brief Title: 18F-NaF Uptake and Aortic Stenosis Progression
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Seoul St. Mary's Hospital (Other)
Responsible Party: Principal Investigator, Ho-Joong Youn, Professor, Seoul St. Mary's Hospital
Other Study IDs: NAFAS
Record Dates: First submitted 2016-04-11; First posted 2016-04-15 (Estimated); Last update posted 2016-04-15 (Estimated); Status verified 2016-04

CONDITIONS: Aortic Stenosis
MeSH Terms: conditions — Aortic Valve Stenosis

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Imaging test: 18F-NaF PET/CT — 18F-NaF PET/CT as an imaging test

SUMMARY:
This study aims to evaluate whether baseline 18F-sodium fluoride uptake activity at aortic valve could predict aortic stenosis progression in moderate aortic stenosis.

Patients with moderate aortic stenosis are enrolled and underwent baseline evaluation including 18F-sodium fluoride PET/CT. After 1 year, all the participants underwent follow-up echocardiography. The study design is an observational trial. Primary endpoint was a change in mean pressure gradient along the aortic valve as assessed by echocardiography at 1 year. Secondary endpoints include changes in aortic valve area, and symptom occurrence.

DETAILED DESCRIPTION:
Recent studies demonstrated 18F-sodium fluoride (NaF) uptake activity as a marker of early-stage calcification. Although valve calcification could be visualized either by echocardiography or coronary computed tomography, they only reflect the current burden of calcium deposit not the activity of calcium deposit. Limited studies exist regarding the usefulness of 18F-NaF uptake at aortic valve for prediction of stenosis progression.

Patients with moderate aortic stenosis - diagnosed by echocardiography - will be enrolled. Enrolled participants will undergo baseline 18F-NaF PET/CT within 6 weeks of baseline echocardiography and followed up for 1 year. After 1 year, all the participants are required to evaluate the aortic stenosis progression by performing echocardiography.

The objective of the study is to test whether baseline 18F-NaF uptake activity predict AS progression.

ELIGIBILITY:
Inclusion Criteria:

* over 20 years old
* moderate aortic stenosis

Exclusion Criteria:

* age < 20 yrs
* pregnant women

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Diagnosed as "moderate aortic stenosis" by echocardiography
Sampling Method: Probability Sample
Enrollment: 28 (Estimated)
Dates: Start 2016-05; Primary Completion 2017-08 (Estimated); Study Completion 2017-11 (Estimated)

PRIMARY OUTCOMES:
mean PG | AS severity progression after 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Ho-Joong Youn, MD, Principal Investigator — Seoul St. Mary's Hospital

IPD SHARING:
Plan to Share IPD: No